CLINICAL TRIAL: NCT02431598
Title: Randomized, Blinded, Placebo-controlled Crossover Study Assessing Association Between Gadolinium-based Contrast Agent Administration and Transient Dyspnea/Arterial Phase Motion Artifact
Brief Title: Eovist vs. Dotarem Healthy Volunteer MRI
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Duke University (Other)
Collaborators: University of California, San Diego (Other); University of Wisconsin, Madison (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Diagnostic
Other Study IDs: Pro00059192
Record Dates: First submitted 2015-04-28; First posted 2015-05-01 (Estimated); Results first posted 2017-04-14 (Actual); Last update posted 2017-04-14 (Actual); Status verified 2017-03

CONDITIONS: Transient Severe Arterial Phase Motion
MeSH Terms: interventions — gadolinium ethoxybenzyl DTPA; gadoterate meglumine; Sodium Chloride

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (3):
- Eovist (gadoxetate disodium) (Active Comparator): While in the MRI scanner, the subject will receive a clinical dose of Eovist, Dotarem, or normal saline. Each subject will receive all three, in random order, blinded to which agent is received in a given instance.
  Interventions: Drug: gadoxetate disodium
- Dotarem (gadoterate dimeglumine) (Active Comparator): While in the MRI scanner, the subject will receive a clinical dose of Eovist, Dotarem, or normal saline. Each subject will receive all three, in random order, blinded to which agent is received in a given instance.
  Interventions: Drug: gadoterate dimeglumine
- Saline (Active Comparator): While in the MRI scanner, the subject will receive a clinical dose of Eovist, Dotarem, or normal saline. Each subject will receive all three, in random order, blinded to which agent is received in a given instance.
  Interventions: Drug: Saline

INTERVENTIONS:
Drug: gadoxetate disodium
  Other Names: Eovist
  Arms: Eovist (gadoxetate disodium)
Drug: gadoterate dimeglumine
  Other Names: Dotarem
  Arms: Dotarem (gadoterate dimeglumine)
Drug: Saline
  Arms: Saline

SUMMARY:
The purpose of this study is to evaluate changes in volunteer breath-holding capacity in response to gadoxetate disodium (Eovist) administration, compared with saline, and gadoterate dimeglumine (Dotarem). Healthy volunteers will be recruited from three study sites. These subjects will be given three, blinded, randomized injections while undergoing an MRI of their liver and holding their breath. During the scan, the subjects' oxygen saturation and heart rate will be closely monitored. Following the scan, the subjects will complete a questionnaire regarding the breath hold.

ELIGIBILITY:
Inclusion Criteria:

- normal renal function (serum eGFR >60)

Exclusion Criteria:

* renal impairment
* allergy to gadolinium-based contrast
* metallic implanted devices
* claustrophobia
* pregnant and lactating females

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 44 (Actual)
Dates: Start 2015-06; Primary Completion 2015-09 (Actual); Study Completion 2015-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Mustafa Bashir, MD, Principal Investigator — Duke University
Locations (1):
- Duke Medical Center, Durham, North Carolina, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Eovist Crossover to Dotarem Crossover to Saline; Dotarem Crossover to Eovist Crossover to Saline; Eovist Crossover to Saline Crossover to Dotarem; Saline Crossover to Dotarem Crossover to Eovist; Dotarem Crossover to Saline Crossover to Eovist; Saline Crossover to Eovist Crossover to Dotarem: Subjects received the agents in this particular order during their MRI.
Period: Overall Study
Arm/Group | Eovist Crossover to Dotarem Crossover to Saline | Dotarem Crossover to Eovist Crossover to Saline | Eovist Crossover to Saline Crossover to Dotarem | Saline Crossover to Dotarem Crossover to Eovist | Dotarem Crossover to Saline Crossover to Eovist | Saline Crossover to Eovist Crossover to Dotarem
Started | 6 | 9 | 9 | 7 | 7 | 6
Completed | 6 | 9 | 9 | 7 | 7 | 6
Not Completed | 0 | 0 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Arm/Group | Eovistvs vs. Dotarem vs. Saline
Number analyzed (Participants) | 44
Age, Continuous [Mean (Standard Deviation); unit: years] | 32 (7.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 24
  Male | 20
Region of Enrollment [Number; unit: participants]
  United States | 44

OUTCOME MEASURES:

1. Primary Outcome: Subject Breath Hold Capacity, as Measured by Number of Seconds a Subject Can Hold His/Her Breath
Time Frame: following contrast administration, up to 5 minutes
Population: All participants received all three drugs.
Measure: Median (Full Range); unit: seconds
Arm/Group | Eovist (Gadoxetate Disodium) | Dotarem (Gadoterate Dimeglumine) | Saline
Number analyzed (Participants) | 44 | 44 | 44
seconds | 28 [8 to 117] | 38 [23 to 125] | 35 [20 to 108]

2. Primary Outcome: Subject-reported Dyspnea, as Measured by Questionnaire Responses
Description: After each breath-hold, the MRI technologist asked the volunteer through the scanner microphone the following two questions, with responses based on a 5-point scale: A) How difficult was it to hold your breath? (1-Not at all; 5-Very difficult); B) Do you feel short of breath now? (1-Not at all; 5-Very short of breath). Responses were recorded for each breath-hold.
Time Frame: following contrast administration, up to 5 minutes
Measure: Mean (Standard Deviation); unit: units on a scale (1-5)
Groups:
- Eovist (Gadoxetate Disodium): Injection of gadoxetate disodium
- Saline: Injection of normal saline
- Dotarem (Gadoterate Dimeglumine): Injection of gadoterate dimeglumine
Arm/Group | Eovist (Gadoxetate Disodium) | Saline | Dotarem (Gadoterate Dimeglumine)
Number analyzed (Participants) | 44 | 44 | 44
units on a scale (1-5)
  Question A | 2.4 (1.1) | 1.8 (1.1) | 1.7 (1.0)
  Question B | 1.3 (0.6) | 1.1 (0.5) | 1.1 (0.4)

3. Secondary Outcome: O2 Saturation Following Contrast Administration
Time Frame: following contrast administration, up to 5 minutes
Measure: Mean (Standard Deviation); unit: percentage
Arm/Group | Eovist (Gadoxetate Disodium) | Dotarem (Gadoterate Dimeglumine) | Saline
Number analyzed (Participants) | 44 | 44 | 44
percentage | 98 (2) | 98 (2) | 98 (2)

4. Secondary Outcome: Heart Rate Following Contrast Injection
Description: Heart rate following contrast injection
Time Frame: following contrast administration, up to 5 minutes
Measure: Mean (Standard Deviation); unit: beats per minute
Arm/Group | Eovist (Gadoxetate Disodium) | Dotarem (Gadoterate Dimeglumine) | Saline
Number analyzed (Participants) | 44 | 44 | 44
beats per minute | 70 (12) | 70 (12) | 70 (12)

5. Secondary Outcome: Percentage of Participants With Transient Severe Motion (TSM) Based on Presence of Motion Artifacts at Arterial Phase Imaging
Description: Arterial-phase breath-holding duration and motion artifacts after each agent were compared using the Mann-Whitney-U test and the McNemar test.
Time Frame: following contrast administration, up to 5 minutes
Measure: Number; unit: percentage of participants with TSM
Arm/Group | Eovist (Gadoxetate Disodium) | Dotarem (Gadoterate Dimeglumine) | Saline
Number analyzed (Participants) | 44 | 44 | 44
percentage of participants with TSM | 7 | 2 | 0

6. Secondary Outcome: Severity of Motion Artifacts at Arterial Phase Imaging, Measured on a 1-5 Scale
Description: 1. no motion artifact
  2. minimal motion artifact
  3. moderate motion artifact
  4. severe motion artifact
  5. extensive motion artifact
Time Frame: following contrast administration, up to 5 minutes
Measure: Mean (Full Range); unit: scores on a scale
Groups:
- Pre-Contrast Phase: Prior to contrast injection
- Arterial Phase: Imaging obtained during arterial phase
- Portal Venous Phase: Imaging obtained during portal venous phase
- Last Dynamic Phase: Imaging obtained during late dynamic phase
Arm/Group | Pre-Contrast Phase | Arterial Phase | Portal Venous Phase | Last Dynamic Phase
Number analyzed (Participants) | 44 | 44 | 44 | 44
scores on a scale
  Eovist | 2.3 [1 to 5] | 2.7 [1 to 5] | 2.4 [1 to 5] | 2.3 [1 to 5]
  Normal Saline | 2.1 [1 to 5] | 2.3 [1 to 5] | 2.2 [1 to 5] | 2.1 [1 to 5]
  Dotarem | 2.2 [1 to 5] | 2.2 [1 to 5] | 2.3 [1 to 5] | 2.3 [1 to 5]

ADVERSE EVENTS:
Arm/Group | Eovist (Gadoxetate Disodium) | Dotarem (Gadoterate Dimeglumine) | Saline
Serious Adverse Events (participants affected / at risk) | 0/44 | 0/44 | 0/44
Other Adverse Events (participants affected / at risk) | 0/44 | 0/44 | 0/44

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No